CLINICAL TRIAL: NCT03686696
Title: Randomized Evaluation of Beta Blocker and Angiotensin Converting Enzyme Inhibitor (ACEI) /Angiotensin Receptor Blocker (ARB) Treatment in MINOCA Patients.
Brief Title: Randomized Evaluation of Beta Blocker and ACEI/ARB Treatment in MINOCA Patients - MINOCA-BAT
Acronym: MINOCA-BAT
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Low inclusion rate.
Sponsor: Uppsala University (Other)
Collaborators: Karolinska Institutet (Other); Göteborg University (Other); University of Leeds (Other); University of Adelaide (Other); Oslo University Hospital (Other); New York University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: EudraCT number 2018-000889-11
Record Dates: First submitted 2018-09-03; First posted 2018-09-27 (Actual); Last update posted 2023-11-27 (Actual); Status verified 2023-11

CONDITIONS: Myocardial Infarction With Non-obstructive Coronary Arteries
Keywords: Myocardial infarction; Treatment; ACE inhibitors; Angiotensin receptor blockade; Beta blockers
MeSH Terms: conditions — MINOCA; Myocardial Infarction | interventions — Adrenergic beta-Antagonists; Angiotensin-Converting Enzyme Inhibitors; Angiotensin Receptor Antagonists

STUDY DESIGN:
Intervention Model Description: 2 * 2 Factorial Design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- No Beta blocker and no ACEI/ARB (No Intervention): No Beta blocker and no ACEI/ARB
- Beta blocker and ACEI/ARB (Experimental): Beta blocker and either ACE inhibitor or Angiotensin receptor blocker
  Interventions: Drug: Beta blocker; Drug: ACEI; Drug: ARB
- Beta blocker alone (Experimental): Beta blocker alone
  Interventions: Drug: Beta blocker
- ACEI/ARB alone (Experimental): Either ACE inhibitor or Angiotensin receptor blocker alone
  Interventions: Drug: ACEI; Drug: ARB

INTERVENTIONS:
Drug: Beta blocker — Patients randomized to beta-blockade will be administered the assigned treatment during the rest of the hospital stay and receive a prescription for the continued use at discharge. The treating physician is encouraged to aim for target dose or highest tolerable dose for the drug. Patients will be encouraged to continue the use of the randomized treatment following discharge until contraindications.
  Other Names: Beta receptor blocker
  Arms: Beta blocker alone; Beta blocker and ACEI/ARB
Drug: ACEI — Patients randomized to ACE inhibitor will be administered the assigned treatment during the rest of the hospital stay and receive a prescription for the continued use at discharge. The treating physician is encouraged to aim for target dose or highest tolerable dose for the drug. Patients will be encouraged to continue the use of the randomized treatment following discharge until contraindications.
  Other Names: ACE inhibitor
  Arms: ACEI/ARB alone; Beta blocker and ACEI/ARB
Drug: ARB — Patients randomized to Angiotensin receptor blockers will be administered the assigned treatment during the rest of the hospital stay and receive a prescription for the continued use at discharge. The treating physician is encouraged to aim for target dose or highest tolerable dose for the drug. Patients will be encouraged to continue the use of the randomized treatment following discharge until contraindications
  Other Names: Angiotensin receptor blocker
  Arms: ACEI/ARB alone; Beta blocker and ACEI/ARB

SUMMARY:
Myocardial infarction with non-obstructive coronary arteries" (MINOCA) occurs in 5-10% of all patients with AMI. There are neither any randomized clinical trials in MINOCA patients evaluating effects of secondary preventive treatments proven beneficial in patients with classic AMI, nor any treatment guidelines.

The primary objective of this multi-national, multi-center pragmatic randomized clinical trial is to determine whether oral beta-blockade compared to no oral beta-blockade, and whether Angiotensin Converting Enzyme Inhibitors (ACEI/ Angiotensin Receptor Blockers (ARB) compared to no ACEI/ARB, reduce the composite endpoint of death of any cause and readmission because of AMI, ischemic stroke or heart failure in patients discharged with myocardial infarction with non-obstructive coronary artery disease (MINOCA) and with no clinical signs of heart failure and with left ventricular (LV) systolic ejection fraction ≥40%.

DETAILED DESCRIPTION:
Large-scale use of acute coronary angiography has revealed a large portion of AMI without angiographically obstructive (defined as ≥50% diameter stenosis) coronary artery disease (CAD). The term "myocardial infarction with non-obstructive coronary arteries" (MINOCA) has been coined for this entity. MINOCA occurs in 5-10% of all patients with AMI and these patients are younger and more often females compared to patients with AMI and obstructive CAD. The 1-year mortality after MINOCA was found to be 3.5% in the systematic review by Pasupathy et al.. There are no randomized clinical trials in MINOCA patients evaluating effects of secondary preventive treatments proven beneficial in patients with classic AMI. However, in an observational study with propensity score matched comparisons the risk of experiencing a Major Adverse Cardiac Event (MACE) was 18% lower in patients treated with ACEI/ARB compared to no ACEI/ARB; in patients on beta blockers compared to patients not using beta blockers there was a non-significant 14% reduction in MACE.

The primary objective of this multi-national, multi-center pragmatic randomized clinical trial is to determine whether oral beta-blockade compared to no oral beta-blockade, and whether ACEI/ARB compared to no ACEI/ARB, reduce the composite endpoint of death of any cause and readmission because of AMI, ischemic stroke or heart failure in patients discharged with myocardial infarction with non-obstructive coronary artery disease (MINOCA) and with no clinical signs of heart failure and with LV systolic ejection fraction ≥40%.

PRIMARY ENDPOINT: Time to death of any cause or readmission because of myocardial infarction, ischemic stroke or heart failure.

SECONDARY ENDPOINTS:

Time to:

* All-cause mortality
* Cardiovascular mortality
* Readmission because of AMI
* Readmission because of ischemic stroke
* Readmission because of heart failure
* Readmission because of unstable angina pectoris
* Readmission because of atrial fibrillation.

Safety:

Time to readmission because of:

* AV-block II-III, hypotension, syncope or need for pacemaker
* Acute kidney injury
* Ventricular tachycardia/fibrillation

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years.
* A clinical diagnosis of MINOCA within the last 30 days.
* Left ventricular ejection fraction ≥40% measured with echocardiography, MRI or left ventriculography after admission and prior to randomization.
* Written informed consent obtained

Exclusion Criteria:

* Any condition that may influence the patient's ability to comply with study protocol.
* Previous revascularization (CABG or PCI)
* Clinical signs of heart failure
* MRI-proven myocarditis or a strong clinical suspicion of myocarditis or takotsubo as cause of the index event
* Contraindications for Beta blocker treatment
* Contraindications for ACEI and ARB treatment
* Prior use of ACEI, ARB, or Beta blockers, which must continue according to treating physician.
* New indication for Beta blocker or ACEI/ARB treatment other than as secondary prevention according to treating physician
* Ongoing pregnancy or woman of childbearing potential not using adequate contraceptives
* Participation in a trial evaluating a drug known to interact with Beta blockers or ACEI/ARB

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Actual)
Dates: Start 2018-12-16 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-08-22 (Actual)

PRIMARY OUTCOMES:
Time to death of any cause, or time to readmission because of AMI, ischemic stroke or heart failure | Time to event from the date of enrollment through study completion, an average of 4 years.
  A Composite of time to all-cause Death and time to re-admission because of AMI, ischemic stroke or heart failure

SECONDARY OUTCOMES:
a All-cause death b Cardiovascular death c Readmission because of AMI d Readmission because of ischemic stroke e Readmission because of heart failure f Readmission because of unstable angina pectoris g Readmission because of atrial fibrillation. | a All-cause death: Time to event from the date of enrollment through study completion, an average of 4 years.

CONTACTS AND LOCATIONS:
Overall Officials: Bertil Lindahl, Prof, Study Chair — Uppsala University
Locations (32):
- Australia (8):
  - Royal Adelaide Hospital, Adelaide, Sout Australi
  - The Lyell McEwin Hospital, Adelaide
  - The Queen Elizabeth Hospital, Adelaide
  - Gold Coast Hospital, Gold Coast
  - Sunshine Hospital, Melbourne
  - Royal Perth Hospital, Perth
  - Gosford Hospital, Sydney
  - John Hunter Hospital, Sydney
- Auckland University Hospital, Auckland, New Zealand
- Norway (2):
  - Haukeland University Hospital, Bergen
  - Oslo University Hospital, Oslo
- Spain (3):
  - Getafe University Hospital, Getafe
  - C.H.U. Ourense, Ourense
  - C.H. Universitario de Santiago, Santiago de Compostela
- Sweden (18):
  - Mälardalens sjukhus Eskilstuna, Eskilstuna
  - Falu Lasarett, Falun
  - Gävle sjukhus, Gävle
  - Sahlgrenska Universitetssjukhus, Sahlgrenska, Gothenburg
  - Hallands sjukhus, Halmstad
  - Helsingborg Lasarett, Helsingborg
  - Ryhovs sjukhus, Jönköping
  - Centralsjukhuset Karlstad, Karlstad
  - Västmanlands sjukhus Köping, Köping
  - Universitetssjukhuset i Linköping, Linköping
  - Skånes Universitetssjukhus Lund, Lund
  - Skånes universtitetssjukhus Malmö, Malmo
  - Vrinneviesjukhuset, Norrköping
  - Örebro University Hospital, Örebro
  - Danderyd Hospital, Stockholm
  - Söderskjukhuset, Stockholm
  - Akademiska Sjukhuset, Uppsala
  - Västerås Lasarett, Västerås

IPD SHARING:
Plan to Share IPD: Yes
We will make a limited, de-identified set of data available for researchers outside the primary investigators two years after the publication of the primary results of the study. Before data are shared, a data-sharing agreement should be established documenting what data are being shared and how the data can be used. The agreement serves two purposes. First, it protects the agency providing the data, ensuring that the data will not be misused. Second, it prevents miscommunication on the part of the provider of the data and the agency receiving the data by making certain that any questions about data use are discussed. The following items should be covered in the data-sharing agreement:
  * Period of agreement
  * Intended use of the data
  * Constraints on use of the data
  * Data confidentiality
  * Data security
  * Methods of data-sharing
Supporting Information: Study Protocol, SAP

REFERENCES:
- [Derived] Nordenskjold AM, Agewall S, Atar D, Baron T, Beltrame J, Bergstrom O, Erlinge D, Gale CP, Lopez-Pais J, Jernberg T, Johansson P, Ravn-Fisher A, Reynolds HR, Somaratne JB, Tornvall P, Lindahl B. Randomized evaluation of beta blocker and ACE-inhibitor/angiotensin receptor blocker treatment in patients with myocardial infarction with non-obstructive coronary arteries (MINOCA-BAT): Rationale and design. Am Heart J. 2021 Jan;231:96-104. doi: 10.1016/j.ahj.2020.10.059. Epub 2020 Oct 24. PMID 33203618